CLINICAL TRIAL: NCT05240469
Title: A Prospective, Parallel-group, Non-inferiority Study to Compare the Efficacy of an Automated Sperm Selection Method Versus Manual Sperm Selection for ICSI
Brief Title: Automated Sperm Selection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Create Fertility Center (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2395
Record Dates: First submitted 2021-10-15; First posted 2022-02-15 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Infertility
Keywords: In Vitro Fertilization; Embryology; Oocyte; Sperm; Automated Sperm Selection; DNA Fragmentation Index
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard sperm selection (No Intervention): In the control group the oocytes will be injected with sperm that is selected by embryologists using conventional methods in the IVF lab.
- Automated sperm selection (Experimental): The only intervention is the additional sperm selection step using software immediately prior to ICSI.
  Interventions: Device: Automated sperm selection software

INTERVENTIONS:
Device: Automated sperm selection software — The software measures both morphology and motility similar to an embryologist but provides a more accurate and consistent measure of sperm characteristics. Embryologists use their experience to qualitatively judge if an individual sperm is "suitable for injection" based on morphology and motility. Similarly, the software follows a two-step process: firstly, a computer vision algorithm measures characteristics of all sperm in a given field, including motility and morphology; secondly, the software algorithm then uses a set of quantitative criteria to categorize and identify the most developmentally competent sperm with normal characteristics. All the characteristics that the software calculate are defined by the WHO guidelines, and the software does not propose or define new parameters.
  Arms: Automated sperm selection

SUMMARY:
Intracytoplasmic sperm injection (ICSI) is one of the standard clinical treatments for infertility. ICSI involves the injection of a single sperm into an oocyte with a sharp micropipette. Injecting a sperm with DNA fragmentation (i.e., physical breakage of the DNA double strands) into the oocyte deterministically lowers the IVF fertilization rate [1][2] and increases the miscarriage rate [3][4]. Since the invention of ICSI in 1992, single sperm selection in ICSI has been made manually by embryologists, who select sperm by qualitatively choosing sperm with "good" motility and/or morphology based on their empirical experience. This involves significant subjectivity and inconsistency. We have developed a robotic system to select sperm with low sperm DNA fragmentation. Automated sperm selection also eliminates the subjectivity and inconsistency in manual sperm selection. The system consists of a camera to acquire images of sperm and a software to analyze the images. Embryologists select sperm by observing the same sperm characteristics as in the software criteria (e.g., speed etc.), but the software provides a more accurate and quantitative measure of sperm characteristics, thus ensuring the selected sperm have low DNA fragmentation.

DETAILED DESCRIPTION:
Intracytoplasmic sperm injection (ICSI) is one of the standard clinical treatments for infertility. ICSI involves the injection of a single sperm into an oocyte with a sharp micropipette. Injecting a sperm with DNA fragmentation (i.e., physical breakage of the DNA double strands) into the oocyte deterministically lowers the IVF fertilization rate [1][2] and increases the miscarriage rate [3][4]. Patients with high sperm DNA fragmentation suffer from repeated IVF failures [8], causing heavy burdens on families and the healthcare system. Since the invention of ICSI in 1992, single sperm selection in ICSI has been made manually by embryologists, who select sperm by qualitatively choosing sperm with "good" motility and/or morphology based on their empirical experience. This involves significant subjectivity and inconsistency.

We have developed a robotic system to select sperm with low sperm DNA fragmentation. Automated sperm selection also eliminates the subjectivity and inconsistency in manual sperm selection. The system consists of a camera to acquire images of sperm and a software to analyze the images. The software automatically measures the 9 motility parameters (e.g., curvilinear speed, path linearity, etc.) and 11 morphology parameters (e.g., head ellipticity, midpiece width etc.). All these 20 parameters are defined by the WHO guidelines [9]. Embryologists select sperm by observing the same sperm characteristics as in the software criteria (e.g., speed etc.), but the software provides a more accurate and quantitative measure of sperm characteristics, thus ensuring the selected sperm have low DNA fragmentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ICSI
* Female partner between 19-43 years of age using own or donor oocytes

Exclusion Criteria:

* Patients who do not provide informed consent
* Patients with less than 6 mature eggs collected
* Patients undergoing IVF without ICSI
* Morphology <4% normal forms
* 100% immotile sperm
* Cases where surgically-retrieved sperm is used for ICSI

Ages: 19 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 330 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Fertilization rate | 1 day
  Fertilization is defined as the visualization of 2 pronuclear at day 1 post ICSI. The proportion of fertilized eggs for each patient will be calculated as fertilization rate. Each patient's data will be aggregated to calculate the overall fertilization rate for all patients.
Blastocyst formation rate | 5 or 6 days
  The proportion of fertilized embryos classified as blastocysts at day 5 or day 6 of development.
Embryo morphology grade as evaluated by the SART grading system | 5 or 6 days
  The morphology grade (good, fair, poor) for each embryo will be evaluated. Grades for all embryos of each patient will be summarized.

SECONDARY OUTCOMES:
Differences in early embryo cleavage divisions and late developmental (blastocyst) morphokinetics. | 5 or 6 days
  Embryo morphokinetic parameters will be calculated from time-lapse embryo development videos using an EmbryoScope embryo culture system. The evaluated morphokinetic parameters for each embryo include:
  * time of pronuclei formation
  * time of cleavage to a two-cell embryo
  * time of cleavage to a three-cell embryo
  * time of cleavage to a four-cell embryo
  * time of cleavage to a six-cell embryo
  * time of cleavage to a eight-cell embryo
  * time to full blastocyst
Differences in the proportion of euploid and aneuploid embryos between the two groups | 5 or 6 days
  Embryo ploidy will be evaluated by preimplantation genetic testing technique for aneuploidy.
Evaluation of patient demographic and stimulation cycle characteristics for confounding variables. | 5 or 6 days
  We will also compare primary outcome measures (fertilization rate, PGT-A results, blastocyst formation rate, embryo grade) of all embryos in the study (control and study group) to the overall rates in the clinic as a measure of quality assurance of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Sun, PhD, Principal Investigator — University of Toronto
Locations (1):
- CReATe Fertility Centre, Toronto, Ontario, Canada